CLINICAL TRIAL: NCT05984810
Title: A Performance Study of SGM-101, a Fluorochrome-labeled Anti-carcinoembryonic Antigen Monoclonal Antibody for Fluorescence-guided Imaging to Determine Local Extent and Resectability During Surgical Resection of Pancreatic Ductal Adenocarcinoma After Neoadjuvant Treatment
Brief Title: NIR-Fluorescence Guided Surgical Resection of Neoadjuvant Treated Localized Pancreatic Cancer Using SGM-101
Acronym: FLUOPANC-II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); Surgimab (Industry)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Surgical oncologist, Head of Vahrmeijer Research Lab, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P23.018; 2023-000026-28 (EudraCT Number); NL82221.058.23 (Registry Identifier: Toetsingonline)
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Adenocarcinoma
Keywords: Fluorescence Guided Surgery; Pancreatic Ductal Adenocarcinoma; Neoadjuvant therapy; Near-Infrared (NIR) Fluorescence imaging; CEA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 10mg, administered 3-5 days before surgery (Experimental): Drug: SGM-101 Intravenous single injection of the targeted NIR fluorophore SGM-101. This targeted 700nm fluorophore developed by SurgiMab S.A.S., Montpellier, France.
  Device: Intraoperative near-infrared fluorescence imaging Intraoperative imaging will be performed with the following CE-marked near-infrared (NIR) fluorescence imaging system: Quest Spectrum imaging platform (v2/3.0). With a NIR-imaging system a potential fluorescent signal of the tumor can be evaluated. Furthermore, the Quest Spectrum platform will also be used for evaluation of ex-vivo fluorescence of resected tissue on the back table (Back table imaging) and pathology department (ex-vivo imaging), which shall be performed during and after every procedure.
  Interventions: Procedure: Fluorescence-guided surgery using CEA-targeted fluorophore SGM-101

INTERVENTIONS:
Procedure: Fluorescence-guided surgery using CEA-targeted fluorophore SGM-101 — Fluorescence-guided surgery using CEA-targeted fluorophore SGM-101

SUMMARY:
Pancreatic carcinoma has a dismal prognosis at time of diagnosis, due to late onset of clinical symptoms, patients present with advance disease. Complete surgical resection is the only potential curative treatment, however only a small percentage is eligible for upfront total surgical resection due to extension into anatomical related important vascular structures. Neoadjuvant chemo(radio)therapy has become the standard treatment modality for non-primary resectable disease (borderline resectable and locally advanced pancreatic cancer (LAPC)), where subsequent downstaging can make identification of the primary tumor more challenging during surgery. Near-infrared (NIR) fluorescence imaging can aid surgeons by providing real-time visualization of tumors, suspect lymph nodes and vital structures during surgery. Additional intra-operative feedback could possibly reduce the frequency of positive resection margins and increase complete removal of locally spread tumor and involved lymph nodes and could thereby improve patient outcomes as well as overall survival. SGM-101 is a targeted NIR-fluorophore, with specific binding capacity for Carcino Embryonic Antigen (CEA) which is overexpressed on tumor cells in the gastro-intestinal tract, including pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a lethal cancer type and is continuously rising as cause of cancer-related death in the Western World. Despite advances in surgical and systemic treatment, the 5-year overall survival (OS) rate remains approximately 10%. This low survival rate is mostly caused by late detection of disease due to the late onset of symptoms. Therefore, most patients are diagnosed with advanced stage disease: at the time of diagnosis, about 15% of patients has (borderline) resectable ((B)RPC) disease (stage I or II), 35% locally advanced pancreatic cancer (LAPC, stage III), and 50% metastatic disease (stage IV). The resectability of disease is determined by the extent of tumor contact with the superior mesenteric artery, celiac artery, superior mesenteric vein, and portal vein.

Over the last decade, preoperative chemo(radio)therapy has increasingly been used in an attempt to downstage BRPC or LAPC and select patients with more favorable tumor biology for resection, with the aim to reduce the chance for (early) recurrence. In essence, only patients showing regression or stable disease without suspected metastatic disease are considered for surgical exploration. However, preoperative therapy complicates the preoperative radiological staging, because conventional imaging modalities cannot differentiate between vital tumor tissue, inflammation and fibrosis induced by the preoperative chemo(radio)therapy. As a consequence, vascular tumor involvement is often overestimated and also hard to interpret with substantial interobserver variability. Therefore, non-progressive disease following preoperative therapy regarding imaging and tumor markers is usually an indication for surgical exploration to determine whether radical resection is achievable.

During surgical exploration preceding intended tumor resection, the surgeon has to assess the extent of local (vascular) tumor involvement based on preoperative imaging and visual and tactile senses. This visual intraoperative White Light Inspection (WLI) combined with tactile feedback, are the main instruments for guidance and decision-making available to surgeons nowadays. As a result of neoadjuvant therapy the appearance, dimensions, and tactile feedback of the target lesion can be altered, mostly as a result of therapy-induced fibrosis, which complicates the assessment of (local) invasiveness. Surgeons benefit from additional tools that give them real-time directional feedback on local tumor status, which is one of the strengths of optical molecular imaging techniques, like Near-infrared fluorescence (NIRF) imaging. Near-infrared fluorescence (NIRF) imaging is an emerging important intraoperative tool for enhancement of visual contrast and is able to provide real-time guidance in tumor visualization and demarcation. Particularly the use of tumor-specific markers coupled to fluorescent imaging moieties show great promise to improve intraoperative staging and allow more radical cytoreductive surgery if considered resectable.

The compound that will be studied in this trial is SGM-101, a CEA-specific chimeric antibody conjugated with a NIR emitting moiety developed by SurgiMab (Montpellier, France). Anti-CEA monoclonal antibodies have been used in more than 100 clinical studies without any toxicity concerns. In addition, it has been shown that it is possible to link an anti-CEA monoclonal antibody to a near-infrared (NIR) emitting fluorophore. Carcinoembryonic antigen (CEA) is a tumor-specific marker that is highly expressed in a number of tumors of epithelial origin (such as colorectal carcinoma and pancreas carcinoma) while it is minimally expressed in normal adult tissues. CEA, among others like Carbohydrate Antigen 19-9 (CA 19-9) is used as diagnostic and prognostic marker during different stages of malignant pancreatic disease. From a previous study conducted in the LUMC with this compound in patients with (borderline) resectable pancreatic cancer the investigators learned that near-infrared fluorescence imaging of pancreatic tumors using a single dose up to 10mg of the anti-CEA targeted fluorophore SGM-101 is safe, well-tolerated, feasible and effective. It results in specific accumulation of SGM-101 in CEA-expressing primary tumors, peritoneal and liver metastases, allowing real-time identification and guidance using intraoperative fluorescence imaging. Furthermore, CEA expression on the targeted PDAC tissue is expected to be none to minimally influenced by the neoadjuvant treatment, either FOLFIRINOX or a combination of Gemcitabine with or without radiotherapy, as described by previous studies. In addition to experience in pancreatic tumors, there is ample experience from finalized phase-II and ongoing phase-III studies in patient with colorectal carcinoma. A recent study in colorectal cancer patients showed that additional malignant lesions were detected and resected using NIR fluorescence imaging in 6 out of 17 patients (35%). Moreover, an expansion on this study showed no SGM-101 related adverse events up to 15 milligrams in 75 patients. There were no trends or clinically relevant changes in vital signs, ECGs or laboratory parameters reported. Any changes in the laboratory results reported in the follow-up moments were related to the surgical procedure. Best imaging results (according to the tumor to background ratio) were achieved with 10 milligrams injected 3 to 5 days prior to surgery.

This study evaluates the yield of NIR-Fluorescence imaging as additional surgical-tool for visualization and assessment of local extent and resectability status of neoadjuvant treated localized pancreatic tumors, local lymph node-involvement as well as potential distant metastatic disease using a single intravenous dose of 10mg SGM-101.

Main objective: Determination of the performance of SGM-101 as a fluorescent tracer for NIR-Fluorescence-guidance (FLI) during surgical pancreatic resections after neoadjuvant therapy for assessment of (local) tumor extent and delineation of the primary tumor, local lymph nodes and potential distant metastatic disease

Design:

Part A: This is a single-center prospective clinical cohort study in patients with neoadjuvant treated non-primarily resectable ((borderline) resectable and locally advanced) pancreatic cancer undergoing scheduled surgical resection. A total of 20 patients will be prospectively enrolled in this study evaluating the performance of NIR-Fluorescence imaging as an additional surgical-tool for the visualization and determination of the local extent of primary tumor, lymph node-involvement and occult hepatic and peritoneal metastatic disease in patients using a single dose of 10mg of SGM-101. The selected dose is based on the pre-clinical and phase I/II results in patients with pancreatic and colorectal cancer.

Part B: Part B is synchronous to part A, to compare and match the TdEV containing blood samples from patients participating in part A this trial needs 20 healthy donor control blood samples of 30mL to address our exploratory endpoints regarding TdEV's. Therefore in this trial 20 healthy volunteers will be asked to participate as anonymous healthy blood donor of 30mL (3 EDTA tubes) peripheral venous blood for a single visit to donate healthy donor blood. The control samples will be used anonymous and there is no further follow-up or additional study related activities.

Investigational drug: The Investigational Medicinal Product (IMP) used in part A is the injectable conjugate SGM-101 is composed of a chimeric monoclonal antibody specific of CEA, bound to a fluorochrome. SGM-101 is manufactured in compliance with Good Manufacturing Practice (GMP). It is a sterile solution for injection supplied in 4 mL amber glass vial (5 mg/mL; 2,3 mL/vial). A dose of 10 mg SGM-101 will be administered intravenously over 30 minutes 3 to 5 (±4) days prior to surgery.

Imaging system: The Investigational Medical Device (IMD) used in part A is the imaging system that will be used in the study is a dedicated NIRF-camera system from Quest Medical Imaging (Quest Medical Imaging, Olympus Europe) the Quest Spectrum 2/3.0 Platform, that is optimized for measurements in the 700-800nm NIR-spectrum. For this device ample handling-experience for end-users exists at the LUMC, gained from standard-of-care and research activities with intra-operative NIRF-imaging.

ELIGIBILITY:
INCLUSION CRITERIA

Part A: To be eligible for inclusion in this study, patients must meet all of the following criteria:

1. Signed informed consent prior to any study-mandated procedure;
2. Patients aged over 18 years old;
3. Has the ability to communicate well with the Investigator in the Dutch/English language and willing to comply with the study restrictions.
4. Neoadjuvant treated (borderline) resectable or locally advanced pancreatic cancer scheduled for a surgical resection

Part B: To be eligible for inclusion in this study, healthy volunteers must meet all of the following criteria:

1. Signed informed consent prior to any study-mandated procedure;
2. Patients aged over 18 years old;
3. Has the ability to communicate well with the Investigator in the Dutch/English language.

EXCLUSION CRITERIA

Part A: To be eligible for conclusion in this study, patients must meet none of the following criteria:

1. History of clinically significant anaphylactic reactions;
2. Previous administration of SGM-101;
3. Pregnant women, or women giving breast feeding;
4. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.

Part B: To be eligible for conclusion in this study, healthy volunteers must meet none of the following criteria:

1. Previous administration of SGM-101;
2. Pregnant women, or women giving breast feeding;
3. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intra-operative visualization of neoadjuvant treated pancreatic tumors using Near-infrared fluorescence imaging, | Surgery -
  The ability to visualize the primary pancreatic tumor, the local tumor extent and resectability status, with adjacent lymph nodes. As well as potential distant metastatic lesions, using SGM-101 and dedicated NIR-imaging systems. Visualization is measured using the tumor-to-background ratio (TBR) in ex-vivo settings. A tumor-to-background ratio (TBR) of at least ≥1.5 provides sufficient contrast for adequate visualization/delineation and will therefore be used as cut-off value.

SECONDARY OUTCOMES:
Concordance between fluorescent signal and tumor status of resected tissue | Through study completion, an average of 3 months
  Concordance to pathology results with respect to the presence of cancer and the imaging assessment, based on fluorescent signal and the tumor status (incl. degree of CEA-expression) of biopsied or resected tissue, expressed as accuracy (%), sensitivity (%) and specificity (%)
Concordance between fluorescent signal and tumor status of resection margins. | Through study completion, an average of 3 months
  Concordance to pathology results with respect to the presence of cancer and the imaging assessment, based on fluorescent signal and the tumor status (incl. degree of CEA-expression) of biopsied or resected tissue, expressed as accuracy (%), sensitivity (%) and specificity (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No